CLINICAL TRIAL: NCT00321191
Title: Measurement of the Second Gas Effect on Sevoflurane in Anaesthetised Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Austin Health (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 02531
Record Dates: First submitted 2006-05-02; First posted 2006-05-03 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2008-08

CONDITIONS: Anesthesia

ARMS (2):
- N2O (Experimental)
  Interventions: Drug: Administration of N2O
- No N2O (Placebo Comparator)
  Interventions: Drug: No nitrous oxide

INTERVENTIONS:
Drug: No nitrous oxide
  Arms: No N2O
Drug: Administration of N2O
  Arms: N2O

SUMMARY:
This study is investigating the "second gas effect", a phenomenon produced by the uptake of nitrous oxide (N2O) by the lungs, during the course of a typical anaesthetic. The effect is to increase the concentration of other breathed gases in the lung. These include oxygen and volatile anaesthetic agents such as sevoflurane, which are also normally administered along with N2O. We wish to i) measure the magnitude of the second gas effects on both blood and expired concentrations of sevoflurane (Part 1), and ii) see if a demonstrable difference exists between the effects on blood and expired concentrations.

DETAILED DESCRIPTION:
This study is investigating the "second gas effect", a phenomenon produced by the uptake of nitrous oxide (N2O) by the lungs, during the course of a typical anaesthetic. The effect is to increase the concentration of other breathed gases in the lung. These include oxygen and volatile anaesthetic agents such as sevoflurane, which are also normally administered along with N2O.

While the second gas effect has been demonstrated previously, by measuring the concentration of volatile anaesthetic in the expired breath, no study has yet shown that it has a significant effect on the concentrations in the blood. The blood concentration is in fact more important, as it directly determines the concentration of anaesthetic reaching the brain, and therefore the effect on the depth of anaesthesia. The second gas effect on blood concentrations may be more powerful than that on expired concentrations, due to the detrimental effect of anaesthesia on the evenness of distribution of ventilation and blood flow in the lung.

The proposed study will have two parallel components or Parts. We wish to i) measure the magnitude of the second gas effects on both blood and expired concentrations of sevoflurane (Part 1), and ii) see if a demonstrable difference exists between the effects on blood and expired concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery requiring relaxant general anaesthesia with arterial blood pressure monitoring via an arterial line.

Exclusion criteria:

* Patients with moderately or severely impaired respiratory disease (FEV1 < 1.5L, or FVC < 2.0L).
* Patients under 18 years of age.
* Morbidly obese patients: BMI > 30
* Patients unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-05; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Fa/FI sevoflurane in 100% O2 vs in 70% N2O and 30% O2 during 1st 60 min anaesthesia
Change in Fa/FI sevoflurane in 100% O2 vs in 70% N2O and 30% O2 after 60 minutes anaesthesia

SECONDARY OUTCOMES:
Fa/FI and FA/FI for N2O will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Peyton, MD FANZCA, Principal Investigator — Austin Health
Locations (1):
- Austin Hospital, Melbourne, Victoria, Australia